CLINICAL TRIAL: NCT01300793
Title: (RICE) Plus Bortezomib (Velcade) in a Dose-Escalating Fashion for Patients With Relapsed or Primary Refractory Aggressive B-Cell NHL
Brief Title: Study of Standard-Dose Rituximab, Ifosfamide, Carboplatin and Etoposide
Acronym: V-RICE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: closed for low accrual and no data is available.
Sponsor: University of California, San Francisco (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06253
Record Dates: First submitted 2009-09-24; First posted 2011-02-23 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Non-Hodgkin's Lymphoma; B-cell Lymphoma
Keywords: V-RICE; Relapsed NHL; Primary Refractory NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Bortezomib; Rituximab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Velcade (bortezomib), rituximab, ifosfamide, carboplatin, etoposide — Rituximab, 375 mg/m2, IV on day 1 Etoposide, 100 mg/m2, IV on days 2 to 4 Carboplatin, AUC 5 (using the Calvert Formula), IV on day 3 Ifosfamide, 5 g/m2 with Mesna 5 g/m2, CIV over 24 hours beginning D. 3 Bortezomib,1.0mg/m2 starting cohort. Based upon a satisfactory safety profile, additional pts. will be enrolled into the 1.3, 1.5 and 1.7mg/m2 cohorts given IVP over 3 sec. d. 1, 4, 8 & 11 q. 28 days.
  Other Names: Velcade, VP-16, Carboplatin, Rituxan, ifosfamide

SUMMARY:
Primary objective of the study is to determine the maximum tolerated dose (MTD) of bortezomib (Velcade) in combination with rituximab, ifosfamide, carboplatin and etoposide for adult patients with relapsed or refractory aggressive B-cell lymphoma. The secondary objectives are to assess the tolerability and safety, the response rate, rate of autologous stem cell transplant and CD34+ progenitor cell collection and engraftment after treatment with this regimen.

DETAILED DESCRIPTION:
Once subjects are determined to be eligible and informed consent is obtained,patients will be enrolled into a starting dose cohort of 1.0mg/m2. Based upon a satisfactory safety profile, additional patients will be enrolled into the 1.3, 1.5 and 1.7mg/m2 cohorts. Each of these dosing cohorts will only be enrolled if satisfactory safety profiles in each of the lower dosing cohorts are obtained. As the process continues, multiple cohorts will be receiving various dosing regimens simultaneously. If a DLT occurs in ≥2 out of 6 patients at the initial dose level, then 3 more patients will be accrued at dose level -1 (0.7mg/m2).

Bortezomib will be given on days 1 (prior to rituximab) and 4, rituximab 375 mg/m2 on day 1, carboplatin AUC 5 and ifosfamide with mesna, each 5 gm/m2, on day 3 and etoposide 100 mg/ m2/day on days 2, 3 and 4 of a 21-day cycle. They will also receive filgrastim on days 6-13 or pegfilgrastim on day 6. Dose-limiting toxicities (DLT) include any grade 3 or 4 non-hematologic toxicities (except alopecia and grade 3 febrile neutropenia), grade 4 febrile neutropenia (life-threatening sepsis) and grade 4 neutropenia persisting past day 35 or grade 3 or 4 thrombocytopenia persisting past day 35.

If there is a DLT at a given bortezomib dose level, 3 more subjects will be enrolled at that dose; if there are 2 or more DLTs then the MTD will be defined as the previous dose level. If at that dose level, >50% of subjects required bortezomib dose reduction, the MTD will be defined as the next lower dose level. Subjects will continue to be accrued in order to treat a minimum of 10 patients at the MTD.

Those who are candidates for autologous stem cell transplant will have CT scan of the neck, chest, abdomen and pelvis after 2 cycles. Subjects with PD or SD will be taken off study. Those with CR, PR or response not meeting PR criteria will undergo a total of 3 cycles of bortezomib + RICE. After the 3rd cycle of bortezomib + RICE, whole body PET/CT scan and bone marrow biopsy will be obtained.

Subjects who achieve CR or PR will then proceed to stem cell mobilization and collection by a standard regimen, followed by autologous stem cell transplant with a preparative regimen to be determined by the investigator. Those with SD or PD will be taken off study. While the mobilization and ASCT procedures are not part of the phase I protocol, outcomes of ASCT will be followed, including CD34+ progenitor cell collection, clinical response to transplant and survival.

Subjects who are not candidates for autologous stem cell transplant will have CT scan of the neck, chest, abdomen and pelvis after the 2nd and 4th cycles. Those who are responding will continue for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Aggressive B-cell non-Hodgkin lymphoma, CD-20 positive, in first relapse or refractory to first- or second-line chemotherapy (non-platinum)

  * Diffuse large B-cell Lymphoma, Mantle Cell Lymphoma, Follicular Lymphoma (Grade III), Transformed Follicular Lymphoma
  * Prior Rituximab is allowed
  * Prior radiation is allowed
  * Prior autologous stem cell transplant is allowed
* Age 18-70 years
* ECOG performance status 0-2
* HIV seronegative
* No CNS involvement: CSF cytology is required for cases with bone marrow involvement, involvement of 2 or more extranodal sites, presentation in the testes or paranasal sinuses, or if any clinical suspicion of CNS involvement (e.g., cranial nerve deficits)
* Measurable disease on CT scan by international working group response criteria • Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* Subject has a platelet count of less than 75,000.
* Subject has an absolute neutrophil count of less than 1000
* Subject has a calculated or measured creatinine clearance of <60 mL/minute within 14 days before enrollment.
* Subject has grade 2 or greater peripheral neuropathy or grade 1 with pain within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Subject has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Subject has been treated with more than two prior chemotherapy regimens
* Subject has been treated with a platinum-based regimen.
* Subject has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-05; Primary Completion 2011-07 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Determine the MTD of Velcade (bortezomib), Rituximab, Ifosfamide, Carboplatin, Etoposide (V-RICE) for patients with relapsed/primary refractory aggressive B-cell non-Hodgkin's lymphoma (NHL) | 5 years

SECONDARY OUTCOMES:
tolerability and safety, response rate, the amount of peripheral blood CD34+ progenitor cells collected and the rate of engraftment, assess the rate of autologous stem cell transplant | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Kaplan, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Unviersity of California Medical Center, San Francisco, California, United States